CLINICAL TRIAL: NCT07300605
Title: The Effects of Kinesio Taping on the Upper Extremity Motor Function, Pain, General Health and Depression in Acute Stroke Patients: A Randomized Controlled Trial
Brief Title: Kinesio Taping for Upper Extremity Motor Function in Acute Stroke Patients
Acronym: KT-AcuteStroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Havvanur Albayrak, Specialist Physician, Department of Physical Medicine and Rehabilitation, SB Istanbul Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUSOM-IRB-2018/249
Record Dates: First submitted 2025-11-30; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke; Upper Extremity Hemiplegia; Kinesio Taping
Keywords: Kinesio Taping; Stroke Rehabilitation; Upper Extremity Recovery; Brunnstrom Stages; Fugl-Meyer Assessment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two parallel groups: kinesio taping and sham taping.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors were blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (Experimental): Participants received kinesio taping applied to the dorsum of the hand and forearm using standard facilitation techniques with approximately 25% tension, in addition to conventional rehabilitation.
  Interventions: Other: Kinesio Taping
- Sham Taping (Sham Comparator): Participants received sham taping without tension and without crossing joints, mimicking the appearance of kinesio taping but without therapeutic effect, in addition to conventional rehabilitation.
  Interventions: Other: Sham Taping

INTERVENTIONS:
Other: Kinesio Taping — Kinesio tape was applied to the dorsum of the hand with five 1-cm I-strips and one 5-cm I-strip extending toward the forearm, with ~25% stretch. Three applications over approximately 3 weeks.
  Arms: Kinesio Taping
Other: Sham Taping — Sham taping was performed using Y- and I-strips without stretch and without crossing joints. Three applications over approximately 3 weeks.
  Arms: Sham Taping

SUMMARY:
This randomized, controlled clinical trial was conducted to evaluate the effects of kinesio taping on upper extremity motor recovery in patients with acute ischemic stroke who presented with flaccid muscle tone. Twenty-six adults were randomly assigned to either a kinesio taping group or a sham taping group, in addition to receiving standard rehabilitation. Participants were evaluated at baseline, at the end of the 3-week taping period, and at 6 weeks using validated measures of motor function, pain, general health, and depression. The study aimed to determine whether kinesio taping provides additional benefits beyond conventional rehabilitation in improving motor performance of the wrist and hand, reducing pain, and supporting overall functional and emotional well-being in the early phase of stroke recovery.

DETAILED DESCRIPTION:
This prospective, randomized, controlled parallel-group trial investigated the clinical effects of kinesio taping on motor recovery of the upper extremity in patients with acute ischemic stroke. Participants were adults aged 50-80 years, within the first six months after stroke, presenting with Brunnstrom Stage 1 flaccid upper extremity and hand. Individuals with hemorrhagic stroke, prior upper limb surgery, severe shoulder pain, additional neurological conditions, or musculoskeletal complications affecting the upper limb were excluded. All participants received standard rehabilitation, including positioning training, conventional exercises, and splinting as needed.

Participants were randomized (1:1) into a kinesio taping group or a sham taping group. The kinesio taping protocol followed standard facilitation techniques applied to the dorsum of the hand and forearm with appropriate tension, aiming to support finger, wrist, and hand activation. Sham taping was performed without tension and without crossing joints, to avoid therapeutic effect while maintaining participant blinding. Both groups received three taping applications over approximately three weeks.

Outcome measures included Brunnstrom staging, Fugl-Meyer Assessment (upper extremity, wrist, and hand subscales), Visual Analog Scale for hand pain, Health Assessment Questionnaire, and Beck Depression Inventory. Evaluations were performed before treatment, at the end of the 3-week intervention period, and at 6 weeks. Statistical analyses were conducted using standard non-parametric methods for intra- and inter-group comparisons.

The study was designed to determine whether kinesio taping provides additional benefit beyond conventional rehabilitation in facilitating neurophysiological recovery, improving wrist and hand motor function, reducing pain, supporting functional independence, and decreasing depressive symptoms in the acute phase of stroke. No adverse events were observed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50-80 years
* Diagnosis of acute ischemic stroke confirmed by CT or MRI
* Within first 6 months after stroke onset
* Brunnstrom Stage 1 for upper extremity and hand (flaccid muscle tone)
* Sufficient cognitive ability to follow instructions
* Participation in inpatient or outpatient stroke rehabilitation
* Ability to provide informed consent

Exclusion Criteria:

* Hemorrhagic stroke etiology
* Prior upper extremity surgery, fracture, contracture, or heterotopic ossification
* Brachial plexus injury or peripheral nerve lesions
* Additional neurological disorders (e.g., Parkinson's disease, spinal cord injury, polyneuropathy)
* Severe shoulder pain (VAS ≥ 5) that could interfere with assessments
* Significant musculoskeletal disorders affecting the hemiplegic upper extremity
* Uncontrolled comorbidities that prevent participation in rehabilitation
* Inability to complete follow-up assessments

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Wrist, Sitting Position Upper Extremity and Hand Scores | Baseline, Week 3, Week 6
  Fugl Meyer Rating Scale (FMRS) was used to evaluate motor function. This scale was developed to evaluate the patient's sensorimotor recovery after stroke by the Brunnstrom motor healing stages. The scale covers the upper extremity in 3 parts: the shoulder-elbow-forearm, the sitting position in the wrist, the hand; and allows the evaluation of reflex activity, synergy patterns and voluntary movements. It is a reliable method for assessing the severity of post-stroke sensorimotor impairment. The maximum total score for the upper extremity in FMRS is 66.

SECONDARY OUTCOMES:
Change in Brunnstrom Staging (Upper Extremity and Hand) | Baseline, Week 3, Week 6
  Combined assessment of upper extremity and hand motor recovery using the Brunnstrom Staging system (Stages 1-6). Higher stages indicate progressive neurophysiological motor recovery in the shoulder-elbow-forearm and hand components.
Change in Visual Analog Scale (VAS) for Hand Pain | Baseline, Week 3, Week 6
  Pain intensity measured using a 10-cm visual analog scale (0 = no pain, 10 = worst pain). Lower scores indicate reduced hand pain.
Change in Health Assessment Questionnaire (HAQ) Disability Index | Baseline, Week 3, Week 6
  Health Assessment Questionnaire (HAQ) was used for the general health evaluation of the patients. HAQ evaluates the functional ability of the patient in both upper and lower extremities. There are 20 questions in eight functionalities that represent a comprehensive range of functional activities, such as dressing, uplifting, eating, walking, hygiene, access, comprehension, and regular activities. The patient's responses are made on a scale from zero (unobstructed) to three (completely disabled).
Change in Beck Depression Inventory (BDI) Score | Baseline, Week 3, Week 6
  Depressive symptoms measured by the Beck Depression Inventory (0-63). Lower scores indicate reduced depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Havvanur Albayrak, Principal Investigator — Koç University School of Medicine
Locations (1):
- SB Istanbul Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT07300605/Prot_000.pdf